CLINICAL TRIAL: NCT01200238
Title: A Phase II Study of the HSP Inhibitor STA-9090 in Metastatic Ocular Melanoma
Brief Title: STA-9090(Ganetespib) in Metastatic Ocular Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Massachusetts General Hospital (Other); Brigham and Women's Hospital (Other); Synta Pharmaceuticals Corp. (Industry)
Responsible Party: Principal Investigator, F. Stephen Hodi, MD, Melanoma Disease Center Director, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-137
Record Dates: First submitted 2010-09-10; First posted 2010-09-13 (Estimated); Results first posted 2018-06-27 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Ocular Melanoma
Keywords: STA9090; STA-9090; HSP90
MeSH Terms: conditions — Uveal Melanoma | interventions — STA 9090

STUDY DESIGN:
Intervention Model Description: The original dose (Cohort A) was amended based on phase 1 data for safety. Therefore there are 2 separate arms reported.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- STA-9090: Cohort A (Experimental): Cohort A participants received STA-9090 200 mg/m2 given intravenously (IV) over 1 hour once weekly (d1, 8, 15 of a 28 day cycle).
  Participants were treated until evidence of disease progression, unacceptable toxicity, intercurrent illness or withdrawal.
  Interventions: Drug: STA-9090
- STA-9090: Cohort B (Experimental): Cohort B participants received STA-9090 150 mg/m2 given intravenously over 1 hour (IV) twice weekly (d1, 4, 8, 11, 15, 18 of a 28 day cycle).
  Participants were treated until evidence of disease progression, unacceptable toxicity, intercurrent illness or withdrawal.
  Interventions: Drug: STA-9090

INTERVENTIONS:
Drug: STA-9090
  Other Names: Ganetespib

SUMMARY:
STA-9090, a synthetic small molecule, demonstrates significant activity for down-regulating Heat Shock Protein 90 or Hsp90 levels. Hsp90 belongs to a class of molecular chaperone proteins known to be critical regulators of cancer cell proliferation and survival. Preclinical laboratory experiments have shown STA-9090, an Hsp90 inhibitor, could inhibit ocular melanoma cell lines. The primary objective of this trial is to obtain evaluations of STA-9090 efficacy to metastatic ocular melanoma.

DETAILED DESCRIPTION:
Patients with metastatic ocular melanoma have a poor prognosis and very limited standard therapeutic options. The recent discoveries of GNAQ and GNA11 mutations leading to MAPK pathway activation and the over-expression of c-Met generate the hypothesis that inhibition of hsp90 client proteins will provide clinical benefit. This study tests the feasibility and efficacy of hsp90 inhibition in patients with metastatic ocular melanoma. Multiple components of the MAPK pathway (B-Raf, C-Raf, cdk4) in addition to c-Met are client proteins of hsp90 and dependent of active hsp90 for stability. Inhibition of hsp90 should lead to decreased expression of these client proteins.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage IV ocular melanoma
* ECOG Performance status 0, 1, or 2
* 18 years of age or older
* Laboratory values as indicated in the protocol
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation
* Presence of metastatic disease that would be amenable to the required biopsies
* At least one site of measurable disease as defined by at least 1cm in greatest dimension. This site must be different from the sites to be used for biopsy. No prior radiation therapy or directed ablation to the site of measurable disease

Exclusion Criteria:

* Chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Major surgery within 4 weeks prior to first dose of STA-9090
* Minor surgery within 7 days of first dose of STA-9090
* Embolization procedure or ablation procedure to treat tumor within 4 weeks of first dose
* Participants may not be receiving any other investigational agents
* Poor venous access for study drug administration unless patient can use silicone based catheters
* History of brain metastases or of leptomeningeal involvement
* History of allergic reactions or hypersensitivity reactions attributed to compounds of similar chemical or biologic composition to STA-9090
* Baseline QTc > 450 msec or previous history of QT prolongation while taking other medications
* Ventricular ejection fraction (EF) of 55% or less at baseline
* Treatment with chronic immunosuppressants
* Melanoma of cutaneous, mucosal or acral-lentiginous origin or of unknown primary
* Prior treatment with HSP90 inhibitor
* Not willing to undergo biopsy before and after treatment
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Other medications, or severe acute/chronic medical or psychiatric conditions or laboratory abnormality that may increase the risk associated with the study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the participant inappropriate for entry into the study
* Pregnant or breastfeeding women
* Individual with a history of a different malignancy are ineligible except for circumstances outlined in the protocol
* HIV-positive individuals on combination antiretroviral therapy
* History of or current coronary artery disease, myocardial infarction, angina pectoris, angioplasty or coronary bypass surgery
* History of or current uncontrolled dysrhythmias, or requirement for antiarrhythmic medication, or Grade 2 or greater left bundle branch block
* NYHA class II/III/IV congestive heart failure with a history of dyspnea, orthopnea or edema that requires current treatment with angiotensin converting enzyme inhibitors, angiotensin II receptor blockers, beta-blockers or diuretics
* Current or prior radiation therapy to the left hemithorax

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-09-17 (Actual); Primary Completion 2014-10-12 (Actual); Study Completion 2016-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: F. Stephen Hodi, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first and last participants registered to cohort A on September 17, 2010 and June 6, 2011 and to cohort B on December 27, 2011 and May 12, 2014.
Period: Overall Study
Arm/Group | STA-9090: Cohort A | STA-9090: Cohort B
Started | 7 | 10
Completed | 0 | 0
Not Completed | 7 | 10
Not completed — Adverse Event | 2 | 1
Not completed — Progressive Disease | 5 | 8
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of all enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | STA-9090: Cohort A | STA-9090: Cohort B | Total
Number analyzed (Participants) | 7 | 10 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (6.5) | 58.5 (18.4) | 58.0 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 2 | 7 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 10 | 17

OUTCOME MEASURES:

1. Primary Outcome: 4-month Progression Free Survival (PFS) Rate
Description: 4-month PFS rate was defined as the proportion of participants alive, absent progression based on Response Evaluation Criteria In Solid Tumors Criteria (RECIST) and on treatment at 4 months. Per RECIST 1.0 criteria: progressive disease (PD) is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Disease was evaluated radiologically at baseline and every 8 weeks on treatment; Relevant for this endpoint was status at 4 months.
Population: The analysis dataset is comprised of all enrolled participants.
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | STA-9090: Cohort A | STA-9090: Cohort B
Number analyzed (Participants) | 7 | 10
proportion of participants | 0.059 [0.003 to 0.25] | 0.118 [0.021 to 0.326]

2. Primary Outcome: Expression of cMET
Description: To estimate the proportion of patients with greater than 50% decrease in expression of HSP90 client protein c-MET 18-24 hours after administration of STA-9090
Time Frame: Estimated up to 24 hours after administration of STA-9090
Population: There was a problem with the assay and therefore this endpoint was not measured.
Arm/Group | STA-9090: Cohort A | STA-9090: Cohort B
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as achieving partial response (PR) or complete response (CR) based on RECIST 1.0 criteria on treatment. Per RECIST 1.0 for target lesions, CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. CR or PR status required confirmation no earlier than 4 weeks following first documentation. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: Disease was evaluated radiologically at baseline and every 8 weeks on treatment; Median treatment duration was 1.8 months for each cohort [range: cohort A (0.9-12.5), cohort B (0.8-31.7)]. Thus, response on treatment was evaluated up to 31.7 months.
Population: The analysis dataset is comprised of all enrolled participants.
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | STA-9090: Cohort A | STA-9090: Cohort B
Number analyzed (Participants) | 7 | 10
proportion of participants | 0.0 [0.0 to 0.348] | 0.10 [0.005 to 0.394]

4. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is defined as achieving stable disease (SD), partial response (P R) or complete response (CR) based on RECIST 1.0 criteria on treatment. Per RECIST 1.0 for target lesions, CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. CR or PR status required confirmation no earlier than 4 weeks following first documentation. Progressive disease (PD) is at least a 20% increase in the sum LD of target lesions from smallest sum LD as reference or the appearance of one or more new lesions. Stable disease (SD) is neither meeting PR or PD. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions. PR or better response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: Disease was evaluated radiologically at baseline and every 8 weeks on treatment; Median treatment duration was 1.8 months for each cohort [range: cohort A (0.9-12.5), cohort B (0.8-31.7)].Thus, response on treatment was evaluated up to 31.7 months.
Population: The analysis dataset is comprised of all enrolled participants.
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | STA-9090: Cohort A | STA-9090: Cohort B
Number analyzed (Participants) | 7 | 10
proportion of participants | 0.286 [0.054 to 0.659] | 0.30 [0.087 to 0.607]

5. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS based on the Kaplan-Meier method is defined as the duration of time from study entry to documented disease progression (PD) requiring removal from the study or death. Per RECIST 1.0 criteria: progressive disease (PD) is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Participants who did not experience progression were censored at date of last disease evaluation.
Time Frame: Dz was evaluated every 8 weeks on treatment; Imaging was obtained as clinically indicated until off-study; Median (range) on-study duration (months) was cohort A: 8.7 (3.7 to 28.7) and cohort B: 4.5 (1.2 to 36.4 months). Thus, follow-up was up to 36.4m.
Population: The analysis dataset is comprised of all enrolled participants.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | STA-9090: Cohort A | STA-9090: Cohort B
Number analyzed (Participants) | 7 | 10
months | 1.6 [0.8 to 3.5] | 1.8 [0.9 to 7.1]

6. Secondary Outcome: Overall Survival (OS)
Description: OS based on the Kaplan-Meier method is defined as the time from study entry to death or date last known alive.
Time Frame: Survival follow-up occurred every 4 weeks long-term; Median (range) on-study duration (months) was cohort A: 8.7 (3.7 to 28.7) and cohort B: 4.5 (1.2 to 36.4 months).Thus, follow-up was up to 36.4m.
Population: The analysis dataset is comprised of all enrolled participants.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | STA-9090: Cohort A | STA-9090: Cohort B
Number analyzed (Participants) | 7 | 10
months | 8.5 [3.7 to 28.7] | 4.9 [3.2 to 13.0]

7. Secondary Outcome: Grade 3-4 Treatment-Related Toxicity Rate
Description: All grade 3-4 adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAEv4 as reported on case report forms were counted to calculate the proportion of participants experiencing at least one treatment-related grade 3 or 4 AE of any type on treatment.
Time Frame: AE assessment was ongoing from the start of study drug and up to day 30 post-treatment. Mean treatment duration was 1.8 months for each cohort [range: cohort A (0.9-12.5), cohort B (0.8-31.7)). Thus, AEs on treatment were followed up to 31.7 months.
Population: The analysis dataset is comprised of all enrolled participants.
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | STA-9090: Cohort A | STA-9090: Cohort B
Number analyzed (Participants) | 7 | 10
proportion of participants | 0.143 [0.007 to 0.521] | 0.80 [0.493 to .963]

ADVERSE EVENTS:
Time Frame: AE assessment was ongoing from the start of study drug and up to day 30 post-treatment; AEs were assessed for the median treatment duration of 1.8 months for each cohort and up to 12.5m in Cohort A and up to 31.7m in Cohort B and then add the 30 days post-treatment.
Description: Maximum grade toxicity by type was first calculated. Serious AEs were defined as grade 3 or higher events with any treatment-attribution. Other AEs were defined as grade 1 or 2 events with any treatment-attribution.
Arm/Group | STA-9090: Cohort A | STA-9090: Cohort B
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/10
Serious Adverse Events (participants affected / at risk) | 2/7 | 9/10
Other Adverse Events (participants affected / at risk) | 7/7 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | STA-9090: Cohort A (N=7) | STA-9090: Cohort B (N=10)
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2
Alkaline phosphatase increased (Investigations) | 0 | 4
Aspartate aminotransferase increased (Investigations) | 0 | 4
GGT increased (Investigations) | 0 | 1
Lipase increased (Investigations) | 2 | 3
Weight loss (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | STA-9090: Cohort A (N=7) | STA-9090: Cohort B (N=10)
Anemia (Blood and lymphatic system disorders) | 1 | 3
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 3
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 | 1
Blurred vision (Eye disorders) | 1 | 1
Eye pain (Eye disorders) | 0 | 1
Floaters (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 4
Anal hemorrhage (Gastrointestinal disorders) | 0 | 1
Anal mucositis (Gastrointestinal disorders) | 0 | 1
Bloating (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 2 | 4
Diarrhea (Gastrointestinal disorders) | 5 | 9
Dry mouth (Gastrointestinal disorders) | 0 | 2
Duodenal hemorrhage (Gastrointestinal disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Esophagitis (Gastrointestinal disorders) | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 1 | 1
Ileal fistula (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 7
Oral pain (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 6
Chills (General disorders) | 0 | 1
Edema limbs (General disorders) | 0 | 1
Fatigue (General disorders) | 4 | 7
Fever (General disorders) | 0 | 2
General disorders and administration site conditions - Other, specify (General disorders) | 0 | 1
Infusion related reaction (General disorders) | 1 | 1
Injection site reaction (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 1
Pain (General disorders) | 4 | 2
Allergic reaction (Immune system disorders) | 1 | 0
Abdominal infection (Infections and infestations) | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 2
Bruising (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 5
Alkaline phosphatase increased (Investigations) | 1 | 5
Aspartate aminotransferase increased (Investigations) | 2 | 5
CPK increased (Investigations) | 0 | 2
Creatinine increased (Investigations) | 0 | 1
Hemoglobin increased (Investigations) | 0 | 1
Lipase increased (Investigations) | 0 | 2
Neutrophil count decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 2
Serum amylase increased (Investigations) | 2 | 2
Weight loss (Investigations) | 1 | 5
White blood cell decreased (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 9
Dehydration (Metabolism and nutrition disorders) | 1 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 3
Hyponatremia (Metabolism and nutrition disorders) | 0 | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2
Dysgeusia (Nervous system disorders) | 0 | 1
Dysphasia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 5
Nervous system disorders - Other, specify (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 2
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 4
Suicidal ideation (Psychiatric disorders) | 1 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 1
Perineal pain (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 2
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 | 3
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 | 1
Flushing (Vascular disorders) | 0 | 1
Hot flashes (Vascular disorders) | 0 | 2
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Vascular disorders - Other, specify (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The study was terminated early due to slow accrual and competing trials.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No